CLINICAL TRIAL: NCT05161390
Title: A Phase I/II , Open, Multicentre, Dose-escalation and Expansion Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Immunogenicity and Antitumour Activity of LM-302 in Patients With CLDN18.2 Positive Advanced Solid Tumours
Brief Title: Study of LM-302 in Patients With Advance Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: LaNova Medicines Zhejiang Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: LaNova Medicines Limited (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LM302-01-102
Record Dates: First submitted 2021-12-05; First posted 2021-12-17 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LM-302 Dose Escalation at different dose levels (Experimental): LM-302 Dose Escalation. 6 dose levels were pre-defined, and the initial accelerated titration followed by the i3+3 design was adopted during phase I.
  Interventions: Drug: LM-302 Injection
- LM-302(RP2D) Dose Expansion (Experimental): LM-302 Dose Expansion, RP2D will be selected for dose expansion, with the aim to further evaluate the preliminary anti-tumor activity, safety and tolerability, etc.
  Interventions: Drug: LM-302 Injection

INTERVENTIONS:
Drug: LM-302 Injection — LM-302 Injection with dose escalation stage of different dose levels, as well as dose expansion stage with recommended dose level from dose escalation stage.

SUMMARY:
A Phase I/II Study of LM-302 in Patients with CLDN18.2-Positive Advanced Solid Tumors

DETAILED DESCRIPTION:
A Phase I/II, First-in-Human, Open-Label, Dose Escalation and Expansion Study of LM-302 in Patients with CLDN18.2-Positive Advanced Solid Tumors The study includes phase I (dose escalation) to determine MTD/RP2D and phase II (dose expansion) to assess the preliminary anti-tumor activity, etc..

ELIGIBILITY:
Inclusion Criteria:

Subjects will be enrolled into the study only if they meet all of the following inclusion criteria:

1. Subjects who are fully informed of the purpose, nature, method and possible adverse reactions of the study, and are willing to participate in the study and sign the informed consent document prior to any procedure;
2. Aged between 18 to 80 years old, male or female when sign the Informed consent form (ICF);
3. ECOG score 0-1;
4. Life expectancy ≥ 3 months;
5. Subjects have histological or cytological confirmation of advanced solid tumors, and are intolerable for available standard therapy, or there is no available standard therapy;
6. Claudin18.2(CLDN18.2) status will be tested by immunohistochemistry (IHC) by central lab, the result must be positive;
7. At least one evaluable lesion for phase I and one measurable lesion for phase II according to RECIST v1.1;
8. Subjects must have the following organ and marrow function in laboratory tests within 7 days prior to the first dose;
9. Subjects who are able to well communicate with investigators as well as understand and adhere to the requirements of this study.

Exclusion Criteria:

Subjects will be excluded from the study, if they meet any of the following criteria:

1. Participate in any other clinical trial within 28 days prior to 1st dosing of LM-302;
2. Subjects with anti-tumor treatment within 21 days prior to 1st dosing of LM-302, including radiotherapy, chemotherapy, biotherapy, endocrine therapy and immunotherapy, etc.
3. Any adverse event from prior anti-tumor therapy has not yet recovered to ≤grade 1 of CTCAE v5.0;
4. Peripheral sensory or motor neuropathy ≥ grade 2;
5. Subjects with uncontrolled tumor-related pain;
6. Subjects with known central meningeal metastasis;
7. Subjects with known brain metastasis, stable brain metastasis judged by investigator can be included;
8. Subjects with uncontrolled third interstitial effusion judged by the investigator to be unsuitable for inclusion;
9. Subjects with known antibody drug allergy ≥ grade 3;
10. Subjects who have received the treatment with ADCs targeting to CLDN18.2;
11. Subjects who were intolerable to the treatment with MMAE based ADCs or anti-CLDN18.2 antibodies are not eligible;
12. Administrate strong inhibitors/strong inducers of CYP3A4 within 14 days prior to 1st dosing of LM-302;
13. Use of any live vaccines within 28 days prior to 1st dosing of LM-302;
14. Subjects with the history of interstitial lung disease or drug-induced interstitial lung disease/pneumonitis;
15. Subjects who are taking therapeutic doses of anticoagulants such as heparin or vitamin K antagonists (except preventive treatment at a stable dose);
16. Uncontrolled persistent and recurrent vomiting (e.g. due to gastric outlet obstruction);
17. Subjects with uncontrolled/severe gastrointestinal hemorrhage, or ulcer within 28 days prior to 1st dosing of LM-302;
18. Subjects who have received surgical or interventional treatment within 28 days prior to 1st dosing LM-302, with the exception for tumor biopsy,puncture, etc.;
19. (Limited PhaseⅡ dose expansion)Subjects who have another active malignancy which is likely to require treatment, and have the history of another malignancy within 2 years before the 1st dosing LM-302;
20. Subjects who have severe cardiovascular disease;
21. Subjects who have uncontrolled or severe illness, including but not limited to ongoing or active infection requiring antibiotics administration;
22. Subjects who have a history of immunodeficiency disease, including other acquired or congenital immunodeficiency diseases, or organ transplantation, or allogeneic bone marrow transplantation, or autologous hematopoietic stem cell transplantation;
23. HIV infection, active HBV and HCV infection;
24. Child-bearing potential female who have positive results in pregnancy test before the 1st dosing LM-302 or are lactating;
25. Subjects who have psychiatric illness or social situations that would preclude study compliance;
26. Subject who is determined as not eligible to participate in this study by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2021-11-26 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | Cycle 1 of each cohort. Duration of one cycle is 21 days
  DLT is defined as a toxicity (adverse event at least possibly related to LM302) occurring during the DLT observation period
Adverse Events and Serious Adverse Events | From signing the ICF until 28 days after EOT or accept other anti-cancer therapy
  The safety profile of LM-302 will be assessed by monitoring the adverse events (AE) per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0
Recommended Phase II Dose (RP2D) | up to 21 days following first dose
  The RP2D will be determined during the dose expansion stage of the study. RP2D will be determined using available safety and efficacy data
Maximum Tolerated Dose (MTD) | up to 21 days following first dose
  The MTD is defined as the dose of which the toxicity rate during the DLT observation period (21 days after the first administration in cycle 1 on day 1).

SECONDARY OUTCOMES:
Area under plasma concentration vs time curve (AUC) for LM-302 | Up to finished cycle 5 (each cycle is 21 days)
  changes in AUC over time in participants with LM-302

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, Principal Investigator — Shanghai East Hospital; Wei Shen, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine; Yuping Sun, Principal Investigator — Shandong Province Cancer Hospital; Yanqiao Zhang, Principal Investigator — The Second Affiliated Hospital of Harbin Medical University; Jianping Xiong, Principal Investigator — The First Affiliated Hospital of Nanchang University; Wenhui Lou, Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China